CLINICAL TRIAL: NCT01529177
Title: Metformin for the Treatment of Unexplained Oligozspermia and Azoospermia
Brief Title: Metformin for the Treatment of Unexplained Oligozspermia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Egyptian IVF-ET Center (Other)
Responsible Party: Principal Investigator, Ragaa Mansour, Director, The Egyptian IVF-ET Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: metformin for spermatogenesis
Record Dates: First submitted 2012-02-04; First posted 2012-02-08 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Infertility
Keywords: Metformin; Insulin resistance; male infertility; unexplained Oligozspermia; Clomiphene citrate; Unexplained azoospermia
MeSH Terms: conditions — Infertility; Insulin Resistance; Infertility, Male | interventions — Metformin; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin / clomid / hCG (Experimental): Metformin 1000 mg orally to be given daily for one week then twice daily for 2 weeks then 3 times daily for 6 months.
  After 3 months from starting metformin the participant will receive 2 more medications in addition to metformin:
  Clomid 50 mg orally per day and 5000 IU human chorionic gonadotrophin (hCG ) IM once per week for three months.
  Interventions: Drug: Metformin / clomid / hCG
- Clomid / hCG (Experimental): Clomid 50 mg per day will be administered orally and human chorionic gonadotrophin ( choriomon ) 5000 IU will be administered IM once per week. Both medications will be given for 6 month.
  Interventions: Drug: Clomiphene citrate / hCG

INTERVENTIONS:
Drug: Metformin / clomid / hCG — Metformin 1000 mg daily for a week then twice daily for 2 weeks then 3 tomes daily for 6 months.
  Other Names: Glucophage / clomiphene citrate / choriomon
  Arms: Metformin / clomid / hCG
Drug: Clomiphene citrate / hCG — Clomiphene citrate 50 mg daily for one month, then twice daily for 2 months then 3 times per day for 3 months.
  Other Names: Clomid / choriomon
  Arms: Clomid / hCG

SUMMARY:
Insulin resistance (IR) in men may be the underlying pathogenesis for metabolic abnormalities and chronic hypospermatogenesis similar to women with polycystic ovarian disease (PCOD). Infertile men with unexplained infertility and IR may benefit from treatment with metformin.

DETAILED DESCRIPTION:
Recently insulin resistance (IR) has been recognized as the underlying pathogenesis of chronic anovulation, hyperandrogenism, and metabolic abnormalities associated with PCOD in women. IR could be the underlying pathogenesis of chronic hypospermatogenesis leading to oligospermia and azoospermia associated with other metabolic abnormalities in men. Metformin has proven as an effective medication for not only IR but several other aspects of the PCOD including reproductive abnormalities. Therefore, insulin sensitizers, particularly metformin can be introduced as a pharmaceutical option for unexplained oligozoospermia and azoospermia associated with insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* oligospermia ( < 10 million per mil-litter )
* normal FSH
* high insulin

Exclusion Criteria:

* abnormal karyotype
* obstructive azoospermia

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-09 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
sperm count | 6 months
  semen analysis before the start of metformin and then every month for 6 months

SECONDARY OUTCOMES:
abnormal forms of spermatozoa | 6 months
  semen analysis before the start of metformin and then every month for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ragaa mansour, MD,PhD, Principal Investigator — The Egyptian IVF-ET Center
Locations (1):
- The Egyptian IVF-ET center, Cairo, Cairo Governorate, Egypt